CLINICAL TRIAL: NCT04232722
Title: An Exploratory Study Evaluating the Efficacy, Safety, and Pharmacokinetics of Sorafenib Combined With Realgar-Indigo Naturalis Formula (RIF) in in Treating Patients With Recurrent Hepatocellular Carcinoma After Liver Transplantation
Brief Title: Sorafenib Combined With Arsenical in Treating Patients With Recurrent HCC After Liver Transplantation
Acronym: HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISLD6
Record Dates: First submitted 2020-01-01; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: HCC
MeSH Terms: interventions — Arsenicals; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sorafenib + arsenical (Experimental): After enrollment, the patients received oral treatment at sorafenib 200mg bid continuous and realgar-indigo naturalis formula preparation at 60mg/kg tid p.o, d1-14, q4w
  Interventions: Drug: Arsenicals

INTERVENTIONS:
Drug: Arsenicals — As4 S4
  Other Names: sorafenib

SUMMARY:
To analyze the safety, efficacy and pharmacokinetic characteristics of sorafenib combined with compound huangdai tablets in patients with recurrent hepatocellular carcinoma after liver transplantation

DETAILED DESCRIPTION:
Background: postoperative recurrence after liver transplantation is a global problem, and there is no standard treatment model for postoperative recurrence. Objective: to select patients diagnosed with hepatocellular carcinoma (HCC) after liver transplantation and unable to receive local treatment, and to give sorafenib combined with realgar-indigo naturalis formula until the disease progression or the patient die or is lost to follow-up. To analyze the safety, efficacy and pharmacokinetic characteristics of sorafenib combined with compound huangdai tablets in patients with recurrent hepatocellular carcinoma after liver transplantation

ELIGIBILITY:
Inclusion Criteria:

* aged 18-75 (inclusive), male or female;
* recurrence of HCC after liver transplantation;
* grade C according to the Barcelona liver cancer classification criteria (BCLC) or grade B not suitable for local treatment/progression of local treatment
* according to RECIST1.1, there was at least one target lesion that could be stably evaluated, defined as: longest diameter of non-lymph node lesion ≥10mm, or shortest diameter of lymph node lesion ≥15mm; The intrahepatic lesions required enhanced arterial development
* expected survival more than 12 weeks;
* child-pugh score ≤7;
* ECOG score 0-1;
* if the subject is HBsAg positive or HBcAb positive, hbv-dna < 200 IU/ml should be satisfied. HBsAg positive subjects must receive antiviral therapy in accordance with the 2015 guidelines for the prevention and treatment of chronic hepatitis B.
* subject should meet the following test results before screening and pretreatment (at baseline). If abnormal laboratory tests do not meet the following criteria, the subjects are allowed to re-examine within one week. If they still do not meet the criteria, the screening will be considered a failure: A. Blood routine (no blood transfusion, platelet transfusion, cell growth factor (except recombinant erythropoietin) and other supportive treatments should be performed within 7 days before the test) : WBC ≥ 2.5×109/L; Platelet count (PLT) ≥60×109/L; Hemoglobin (Hb) ≥ 9.0g /dL; B. Blood biochemistry: serum albumin (Alb) ≥30 g/L; The clearance rate of endogenous creatinine was ≥50 mL/min (Cockcroft -Gault formula was used). Alanine aminotransferase (ALT) ≤5× upper limit of normal value (ULN); Aspartate aminotransferase (AST) ≤5×ULN; Alkaline phosphatase ≤5×ULN; Total bilirubin ≤2×ULN; C. Prothrombin time (PT) : prothrombin time extension ≤ 4 s;
* women of child-bearing age must undergo a serum pregnancy test within the screening period and 14 days prior to the initiation of the study drug, with negative results, and be willing to use reliable methods of contraception during the test period; Male subjects whose partners are women of child-bearing age should be sterilized or agree to use reliable methods of contraception during the trial;
* be able to understand and sign the informed consent.

Exclusion Criteria:

* participate in other clinical trials or use other research drugs or devices within 4 weeks of the first treatment.
* pregnant or breastfeeding women;
* positive for human immunodeficiency virus (HIV) antibody, treponema pallidum antibody or hepatitis C virus (HCV-RNA) antibody;
* any uncontrolled active infection, including but not limited to subjects with active tuberculosis;
* previous or present hepatic encephalopathy;
* the presence of clinically significant ascites is defined as the ascites that are positive on physical examination or that need to be controlled by intervention therapy (for example, puncture or drug therapy, etc.).
* imaging results: the proportion of liver replaced by tumor was ≥50%, and the main portal vein tumor thrombus or tumor thrombus invaded mesenteric vein/inferior vena cava;
* adverse reactions caused by previous treatment did not return to the standard term for adverse events (CTCAE) ≤1, except hair loss and other tolerable events judged by researchers;
* subjects who currently have unstable or active ulcers, gastrointestinal bleeding, or intolerance to proton pump inhibitors;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | Through the study peirod, for 18 months
  objective response rate

SECONDARY OUTCOMES:
PFS | Through the study peirod, for 18 months
  progression-free survival
DCR | Through the study peirod, for 18 months
  disease control rate
OS | Through the study peirod, for 18 months
  overall survival
Safty | Through the study peirod, for 18 months
  adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No